CLINICAL TRIAL: NCT00195637
Title: Pilot Study of the Use of Intravenous Immune Globulin in Hereditary Inclusion Body Myopathy
Brief Title: Intravenous Immune Globulin to Treat Hereditary Inclusion Body Myopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050236; 05-HG-0236
Record Dates: First submitted 2005-09-18; First posted 2005-09-19 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2018-05-22

CONDITIONS: Hereditary Inclusion Body Myopathy
Keywords: GNE Gene; Alpha-Dystroglycan; Sialic Acid; Glycosylation; Dystroglycanopathy; Hereditary Inclusion Body Myopathy; Immune Globulin; HIBM
MeSH Terms: conditions — Distal myopathy, Nonaka type | interventions — Immunoglobulins

INTERVENTIONS:
Drug: Immune Globulin

SUMMARY:
This study will evaluate patients with Hereditary Inclusion Body Myopathy (HIBM) and examine the effects of immune globulin (IG) treatment on muscle and muscle function. HIBM is a progressive neuromuscular disease that begins in early adulthood, primarily affecting limb muscles. It results from mutations of the gene that is responsible for producing sialic acid, a sugar normally found on the surface of certain proteins, including alpha-dystroglycan, which is involved in muscle function. Some patients with HIBM have decreased sialic acid on the alpha-dystroglycan protein, which may be the cause of their muscle weakness. IG is a protein in the blood that carries a large amount of sialic acid. This study will administer IG to patients with HIBM and determine if the sialic acid in IG is taken up by muscle cells in these patients and if it can restore some of their muscle function.

Four patients with HIBM will be admitted to this study at the NIH Clinical Center for evaluation and IG treatment. The evaluation lasts about 1 month. After completing baseline studies (see below), patients receive two intravenous doses of immune globulin (on days 6 and 7), followed by measurement of muscle strength 2 days later (day 9). They receive additional IG infusions on days 13, 20, and 27. A final set of tests is performed on day 29. Patients may leave the hospital on pass when no studies are being done.

A patient's initial evaluation includes:

* History and physical examination, neurological examination, eye examination
* 24-hour urine collection
* Blood tests on two separate days
* Photographs showing the extent of muscle affected
* Chest x-ray, electrocardiogram (EKG), and echocardiogram
* Two muscle biopsies, one before and one after the IG treatments. For this procedure, a small sample of muscle tissue is surgically removed for examination under the microscope.
* Muscle strength and endurance testing, including the following:

The patient uses pulleys attached to machines that measure the strength of 24 different muscle groups

The patient walks for 6 minutes and performs exercises

To evaluate swallowing, the patient swallows a thick substance called barium

The patient's tongue strength is measured using a specialized instrument.

-Magnetic resonance imaging (MRI) of the muscles of the thigh or calf: MRI uses a magnetic field and radio waves to produce detailed pictures of organs and tissues. During the scan, the subject lies on a table in a narrow cylinder containing a magnetic field, wearing ear plugs to muffle loud noises that occur with electrical switching of the magnetic fields. He or she can speak with a staff member via an intercom system at all times during the procedure.

The neurological and muscle strength and endurance evaluations are repeated on study days 9 and 29.

DETAILED DESCRIPTION:
Hereditary Inclusion Body Myopathy (HIBM) is an autosomal recessive neuromuscular disorder with onset in early adulthood and progressive muscle weakness leading to death within 2-3 decades. The causative gene, GNE, codes for the bifunctional enzyme UDP N-acetylglucosamine 2-epimerase/N-acetylmannosamine kinase; mutations on both GNE alleles, in either or both the epimerase and kinase domains, can result in HIBM. Members of an Iranian-Jewish isolate are homozygous for a specific kinase domain mutation. The epimerase and kinase enzymes catalyze the first and second, rate-limiting steps in the synthesis of sialic acid, also called N-acetylneuraminic acid. This charged sugar provides the terminal carbohydrate on a variety of N-linked and O-linked glycoproteins that mediate cell-cell and protein-protein interactions. The cells of HIBM patients produce reduced amounts of free sialic acid, as evidenced by decreased sialylation of glycoproteins, including a critical muscle protein called alpha-dystroglycan (alpha-DG). This protein, decorated with O-mannosyl glycans containing a terminal sialic acid, is part of the dystrophin-glycoprotein complex responsible for linking the inside of muscle cells with the extracellular matrix. In HIBM, improper sialylation of alpha-DG, due to decreased sialic acid synthesis, is considered to impair the interactions of alpha-DG with its protein ligands, resulting in gradual deterioration of muscle cells. In this open-label pilot study, we propose to provide free sialic acid to muscle cells of HIBM patients by intravenous infusions of immune globulin (IvIg), a glycoprotein that contains 8 microlitermoles of sialic acid per gram and that has a proven safety profile as an FDA-approved drug. Four subjects will be treated - two homozygous for the Iranian Jewish kinase domain mutation, and two with at least one epimerase domain mutation. IvIg will be given as a loading dose of 1 gram per kilogram body weight on two consecutive days, followed each of the next 3 weeks by maintenance doses of 400 milligram per kilogram body weight. This should maintain the serum immune globulin level high enough to achieve continuous breakdown of large amounts of the glycoprotein, providing free sialic acid to the blood, scavenger cells and, we hope, muscle cells. Muscle biopsies and strength testing will be performed before and after the infusions. The primary clinical outcome parameter will be muscle strength, gauged mechanically by Quantitative Muscle Testing and manually by physical examination performed by a neurologist. Secondary outcome parameters will employ the 6-minute walk test, grip strength, tongue strength, swallowing duration, and the Human Activity Profile questionnaire. Staining of muscle beta-DG for sialic acid on O-mannosyl glycans will provide a histological outcome parameter. An improvement in muscle strength or alpha-DG sialylation will prompt a controlled trial of the efficacy of this treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-70 years, either gender
* Diagnosis of HIBM based upon a consistent clinical course plus either convincing muscle histology or identification of GNE gene mutations
* Ability to travel to the NIH Clinical Research Center for admissions

EXCLUSION CRITERIA:

* Age less than18 or greater than 70, pregnancy
* Previous adverse reaction to IvIg that did not resolve with acetaminophen or benadryl treatment
* History of myocardial infarction, stroke, or kidney disease
* Psychiatric illness or neurological disease that interferes with compliance or communication with health care personnel
* Current malignancy
* Uncontrolled hypertension (blood pressure greater than180 systolic or greater than 95 diastolic)
* Electrocardiogram changes indicative of myocardial infarction, arrhythmia, tachycardia, bradycardia, left bundle branch block
* Chest radiographic abnormalities, including an infiltrate, mass, congestive heart failure, embolism, atelectasis
* Serum potassium less than 3.0 mEq/L
* Serum creatinine greater than 2.0 mg/dL
* SGPT or SGOT greater than 70 U/L
* Hemoglobin less than 10.0 g/dL
* Platelets less than100 k/mm(3)
* WBC less than 3.0 k/microliters
* ESR greater than100 mm/h

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-09-16; Primary Completion 2006-07-03 (Actual); Study Completion 2006-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Griggs RC, Askanas V, DiMauro S, Engel A, Karpati G, Mendell JR, Rowland LP. Inclusion body myositis and myopathies. Ann Neurol. 1995 Nov;38(5):705-13. doi: 10.1002/ana.410380504. No abstract available. PMID 7486861
- [Background] Sadeh M, Gadoth N, Hadar H, Ben-David E. Vacuolar myopathy sparing the quadriceps. Brain. 1993 Feb;116 ( Pt 1):217-32. doi: 10.1093/brain/116.1.217. PMID 8453459
- [Background] Sivakumar K, Dalakas MC. The spectrum of familial inclusion body myopathies in 13 families and a description of a quadriceps-sparing phenotype in non-Iranian Jews. Neurology. 1996 Oct;47(4):977-84. doi: 10.1212/wnl.47.4.977. PMID 8857730